CLINICAL TRIAL: NCT05615480
Title: Effect of Controlled Hypotension Guided by Cerebral Oxygen Saturation Monitoring on Postoperative Cognitive Function of Elderly Patients Undergoing Shoulder Arthroscopy
Brief Title: Effect of Cerebral Oxygen Saturation Monitoring on POCD of Elderly Patients Undergoing Shoulder Arthroscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-KY-009-001
Record Dates: First submitted 2022-05-09; First posted 2022-11-14 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2022-05

CONDITIONS: Cerebral Oxygen Saturation; Postoperative Cognitive Function
Keywords: controlled hypotension

STUDY DESIGN:
Intervention Model Description: Recruited patients will be randomly divided into control group and experimental group according to whether cerebral oxygen saturation monitoring was used during the operation. The control group maintain the target blood pressure only according to the controlled hypotension guideline, and the experimental group adjust the controlled hypotension level under the guidance of cerebral oxygen saturation monitoring.
Who Masked: Participant, Outcomes Assessor
Masking Description: In this study, different researchers will be responsible for randomization, anesthesia and visit. A researcher is responsible for assigning random numbers to ensure the randomness of the study groups. Due to the intraoperative monitoring of cerebral oxygen saturation in the experimental group, it is impossible to blind the researchers implementing anesthesia. In order to ensure that the whole study is not affected by subjective factors, the visiting researchers are blinded, who do not know the anesthesia grouping, and are responsible for case enrollment screening, signing informed consent, preoperative and postoperative cognitive function evaluation, postoperative pain evaluation, complications and safety evaluation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group maintain the target blood pressure only according to the controlled hypotension guideline.
- Experimental group (Experimental): The experimental group adjust the controlled hypotension level under the guidance of cerebral oxygen saturation monitoring.
  Interventions: Other: Controlled hypotension guided by cerebral oxygen saturation monitoring

INTERVENTIONS:
Other: Controlled hypotension guided by cerebral oxygen saturation monitoring — In this group, intraoperative monitoring of cerebral oxygen saturation will be used. When the cerebral oxygen saturation decreased by 20% ~ 25% compared with the baseline for 300 seconds without improvement, or the cerebral oxygen saturation decreased by 25% ~ 30% compared with the baseline for 180 seconds without improvement, intervention would be carried out. When the cerebral oxygen saturation decreased by 30% compared with the baseline, immediate intervention would be carried out. The intervention measures were intravenous administration of deoxyepinephrine 50 ~ 100 μg or ephedrine 5 ~ 10mg, which can be administered multiple times until the cerebral oxygen saturation reaches more than 80% of the baseline.
  Arms: Experimental group

SUMMARY:
To observe whether adjusting the level of intraoperative controlled hypotension through cerebral oxygen saturation monitoring can improve postoperative cognitive function(POCD) and reduce postoperative neurological complications, a prospective randomized controlled study method will be used in this study. 400 elderly patients undergoing shoulder arthroscopic surgery under general anesthesia combined with brachial plexus block will be selected. They will be randomly divided into control group and experimental group according to whether cerebral oxygen saturation monitoring was used during the operation. The control group maintain the target blood pressure only according to the controlled hypotension guideline, and the experimental group adjust the controlled hypotension level under the guidance of cerebral oxygen saturation monitoring. The general condition, operation, anesthesia and hospitalization related data of the patients will be recorded.

DETAILED DESCRIPTION:
Cognitive function will be evaluated within 3 days before operation and 3 days, 14 days and 3 months after operation. Delirium and VAS pain score will be evaluated 24 hours after operation. Venous blood will be taken before operation and 24 hours after operation to detect cognitive related markers and inflammatory factors. In addition, 10 blood samples of patients in each group were selected for RNA omics test. One month, six months and 12 months after operation, cognitive function was evaluated by cognitive function telephone questionnaire (TICS-M), and the ability of daily living was evaluated by IDAL. In addition, 20 non-surgical patients were selected for cognitive function evaluation at the same time point as the exercise effect of POCD detection.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective shoulder arthroscopic surgery under general anesthesia combined with brachial plexus block;
* ASA grade ≤ grade III;
* Patients Can communicate normally, can cooperate and complete cognitive function test;
* Patients volunteered and signed informed consent.

Exclusion Criteria:

* BMI < 18 or > 27 kg / m2;
* Previous history of dementia, psychosis or other central nervous system diseases or mental diseases, such as cerebral infarction, stroke, Parkinson's disease, etc;
* Patients taking sedatives or antidepressants;
* Alcoholics or drug addicts;
* Illiteracy, severe hearing or visual impairment;
* Patients with cognitive impairment before operation (MMSE score < 23);
* Patients with peripheral vascular diseases and contraindication of arterial puncture and catheterization;
* Patients unable to carry out long-term follow-up or poor compliance.

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative cognitive dysfunction(POCD) 3 days after operation | 3 days after operation
  The Neuropsychological test, includes: (1) Vocabulary learning; (2) Vocabulary recall; (3) Connection test; (4) Stroop Color word interference; (5) Letter-number coding test.

SECONDARY OUTCOMES:
Incidence of postoperative cognitive dysfunction(POCD) 14 days after operation | 14 days after operation
  The Neuropsychological test, includes: (1) Vocabulary learning; (2) Vocabulary recall; (3) Connection test; (4) Stroop Color word interference; (5) Letter-number coding test.
Incidence of postoperative cognitive dysfunction(POCD) 3 months after operation | 3 months after operation
  The Neuropsychological test, includes: (1) Vocabulary learning; (2) Vocabulary recall; (3) Connection test; (4) Stroop Color word interference; (5) Letter-number coding test.
Expression changes of cognitive function related markers 24 hours after operation | 24 hours after operation
  Patients consented on blood sampling receive marker analysis from blood（S100β、NSE and IL-6).
Hospital stay | through hospitalization period, an average of 15 day
  Hospital stay
Hospital expenses | through hospitalization period, an average of 15 day
  Hospital expenses
Perioperative complications | 1 day (during the surgical period)
  Complications during the surgical period

OTHER OUTCOMES:
Safety outcomes | through study completion, an average of 1 year
  Complications and adverse reactions of patients during the study period

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daiello LA, Racine AM, Yun Gou R, Marcantonio ER, Xie Z, Kunze LJ, Vlassakov KV, Inouye SK, Jones RN, Alsop D, Travison T, Arnold S, Cooper Z, Dickerson B, Fong T, Metzger E, Pascual-Leone A, Schmitt EM, Shafi M, Cavallari M, Dai W, Dillon ST, McElhaney J, Guttmann C, Hshieh T, Kuchel G, Libermann T, Ngo L, Press D, Saczynski J, Vasunilashorn S, O'Connor M, Kimchi E, Strauss J, Wong B, Belkin M, Ayres D, Callery M, Pomposelli F, Wright J, Schermerhorn M, Abrantes T, Albuquerque A, Bertrand S, Brown A, Callahan A, D'Aquila M, Dowal S, Fox M, Gallagher J, Anna Gersten R, Hodara A, Helfand B, Inloes J, Kettell J, Kuczmarska A, Nee J, Nemeth E, Ochsner L, Palihnich K, Parisi K, Puelle M, Rastegar S, Vella M, Xu G, Bryan M, Guess J, Enghorn D, Gross A, Gou Y, Habtemariam D, Isaza I, Kosar C, Rockett C, Tommet D, Gruen T, Ross M, Tasker K, Gee J, Kolanowski A, Pisani M, de Rooij S, Rogers S, Studenski S, Stern Y, Whittemore A, Gottlieb G, Orav J, Sperling R; SAGES Study Group*. Postoperative Delirium and Postoperative Cognitive Dysfunction: Overlap and Divergence. Anesthesiology. 2019 Sep;131(3):477-491. doi: 10.1097/ALN.0000000000002729. PMID 31166241
- [Background] Steinmetz J, Christensen KB, Lund T, Lohse N, Rasmussen LS; ISPOCD Group. Long-term consequences of postoperative cognitive dysfunction. Anesthesiology. 2009 Mar;110(3):548-55. doi: 10.1097/ALN.0b013e318195b569. PMID 19225398
- [Background] Evered LA, Silbert BS, Scott DA, Maruff P, Ames D. Prevalence of Dementia 7.5 Years after Coronary Artery Bypass Graft Surgery. Anesthesiology. 2016 Jul;125(1):62-71. doi: 10.1097/ALN.0000000000001143. PMID 27127919
- [Background] Krenk L, Rasmussen LS, Kehlet H. New insights into the pathophysiology of postoperative cognitive dysfunction. Acta Anaesthesiol Scand. 2010 Sep;54(8):951-6. doi: 10.1111/j.1399-6576.2010.02268.x. Epub 2010 Jul 12. PMID 20626359
- [Background] Moller JT, Cluitmans P, Rasmussen LS, Houx P, Rasmussen H, Canet J, Rabbitt P, Jolles J, Larsen K, Hanning CD, Langeron O, Johnson T, Lauven PM, Kristensen PA, Biedler A, van Beem H, Fraidakis O, Silverstein JH, Beneken JE, Gravenstein JS. Long-term postoperative cognitive dysfunction in the elderly ISPOCD1 study. ISPOCD investigators. International Study of Post-Operative Cognitive Dysfunction. Lancet. 1998 Mar 21;351(9106):857-61. doi: 10.1016/s0140-6736(97)07382-0. PMID 9525362
- [Background] Newman MF, Grocott HP, Mathew JP, White WD, Landolfo K, Reves JG, Laskowitz DT, Mark DB, Blumenthal JA; Neurologic Outcome Research Group and the Cardiothoracic Anesthesia Research Endeavors (CARE) Investigators of the Duke Heart Center. Report of the substudy assessing the impact of neurocognitive function on quality of life 5 years after cardiac surgery. Stroke. 2001 Dec 1;32(12):2874-81. doi: 10.1161/hs1201.099803. PMID 11739990
- [Background] Needham MJ, Webb CE, Bryden DC. Postoperative cognitive dysfunction and dementia: what we need to know and do. Br J Anaesth. 2017 Dec 1;119(suppl_1):i115-i125. doi: 10.1093/bja/aex354. PMID 29161395
- [Background] Tang L, Kazan R, Taddei R, Zaouter C, Cyr S, Hemmerling TM. Reduced cerebral oxygen saturation during thoracic surgery predicts early postoperative cognitive dysfunction. Br J Anaesth. 2012 Apr;108(4):623-9. doi: 10.1093/bja/aer501. Epub 2012 Feb 5. PMID 22311364
- [Background] Kim J, Shim JK, Song JW, Kim EK, Kwak YL. Postoperative Cognitive Dysfunction and the Change of Regional Cerebral Oxygen Saturation in Elderly Patients Undergoing Spinal Surgery. Anesth Analg. 2016 Aug;123(2):436-44. doi: 10.1213/ANE.0000000000001352. PMID 27285000
- [Background] de Tournay-Jette E, Dupuis G, Bherer L, Deschamps A, Cartier R, Denault A. The relationship between cerebral oxygen saturation changes and postoperative cognitive dysfunction in elderly patients after coronary artery bypass graft surgery. J Cardiothorac Vasc Anesth. 2011 Feb;25(1):95-104. doi: 10.1053/j.jvca.2010.03.019. Epub 2010 Jul 22. PMID 20650659
- [Background] Nilsson PM. The J-shaped curve in secondary prevention: shall clinical practice change? Hypertension. 2012 Jan;59(1):8-9. doi: 10.1161/HYPERTENSIONAHA.111.182774. Epub 2011 Nov 7. No abstract available. PMID 22068873
- [Background] Erdem AF, Kayabasoglu G, Tas Tuna A, Palabiyik O, Tomak Y, Beyaz SG. Effect of controlled hypotension on regional cerebral oxygen saturation during rhinoplasty: a prospective study. J Clin Monit Comput. 2016 Oct;30(5):655-60. doi: 10.1007/s10877-015-9768-6. Epub 2015 Sep 10. PMID 26358703
- [Background] Cox RM, Jamgochian GC, Nicholson K, Wong JC, Namdari S, Abboud JA. The effectiveness of cerebral oxygenation monitoring during arthroscopic shoulder surgery in the beach chair position: a randomized blinded study. J Shoulder Elbow Surg. 2018 Apr;27(4):692-700. doi: 10.1016/j.jse.2017.11.004. Epub 2018 Feb 1. PMID 29396097
- [Background] Salazar D, Sears BW, Aghdasi B, Only A, Francois A, Tonino P, Marra G. Cerebral desaturation events during shoulder arthroscopy in the beach chair position: patient risk factors and neurocognitive effects. J Shoulder Elbow Surg. 2013 Sep;22(9):1228-35. doi: 10.1016/j.jse.2012.12.036. Epub 2013 Feb 15. PMID 23415820